CLINICAL TRIAL: NCT03866681
Title: Sirolimus Combined With Low-dose Warfarin for the Treatment of Refractory Classic Paroxysmal Nocturnal Hemoglobinuria ,a Prospective Study
Brief Title: Sirolimus Combined With Low-dose Warfarin for the Treatment of Refractory PNH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Clinical Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hanb
Record Dates: First submitted 2019-02-28; First posted 2019-03-07 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — Sirolimus; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients cohort (Experimental): A total of 40 patients with refractory classic PNH will be included and will be intervened by a combined therapy including sirolimus and low-dose warfarin
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — The dose of sirolimus is adjusted according to monitored serum concentration, maintain Rapamycin concentration ranging from 4 to 10ng/ml.Warfarin was administered orally at a dose of 1mg per day for a year,then gradually reduced to stop.
  Other Names: warfarin

SUMMARY:
Classical paroxysmal nocturnal hemoglobinuria(PNH) is mainly characterized by hemolysis and thrombosis, which reduced patients ' quality of life(QoL) greatly and even lead to death. Glucocorticoids and symptomatic supportive therapy are traditional treatments and the response rate is far from satisfactory. Eculizumab is an effective therapy but it is expensive and not available in China mainland.The investigators aim to explore the efficacy and safety of sirolimus for refractory classic PNH.

DETAILED DESCRIPTION:
Classical paroxysmal nocturnal hemoglobinuria(PNH) is mainly characterized by hemolysis and thrombosis, which reduced patients ' quality of life(QoL) greatly and even lead to death. There is no ideal therapy except for eculizumab, expensive and not available in China mainland. Glucocorticoids and symptomatic supportive therapy are traditional treatments. The response rate is 30%, far from satisfactory. In recent years, T lymphocyte-mediated destruction of normal hematopoietic stem cells have been reported to involve the pathogenesis of PNH, making immunomodulatory drugs be potential effective treatments.

Sirolimus (rapamycin), produced by the bacterium Streptomyces hygroscopicus, is a mammalian target of Rapamycin (mTOR) inhibitor. mTOR is a serine/threonine kinase that regulates cell growth, proliferation, metabolism and survival. It has two interacting complex, mTORC1 and mTORC2. Sirolimus primarily inhibits mTORC1, has been demonstrated for its immunomodulatory effects and ability to improve hematopoietic stem cell function. Recently, sirolimus has been reported to be effective and well tolerated in the treatment of immune-mediated cytopenias, even in multi-immunosuppressants resistant patients. In addition, classical PNH patients have a higher risk of thrombosis especially in refractory ones and it is reasonable to use low-dose warfarin in the management of patients with classic refractory PNH.

In this study, it is anticipated to evaluate the effect of sirolimus combined with low-dose warfarin on patients with refractory classic PNH. The adverse effects and QoL on different time points were documented.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years
* diagnosed with PNH and no thrombosis
* ineffective, relapsed or intolerant to conventional treatment (eg glucocorticoids, • • iron, folic acid, androgen, etc.)
* not available for hematopoietic stem cell transplantation
* ECOG≤2
* agreed to sign the consent forms

Exclusion Criteria:

* severe heart, liver and kidney dysfunction
* combined with thrombotic complications
* people who are pregnant and breastfeeding
* history of other immunosuppressive agents in recent 3 months
* Patients who are not eligible to participate in this trial due to any reason based • • • on the consideration of investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | 2 years
  Hemoglobin in g/L

SECONDARY OUTCOMES:
Short Form 36 items(SF-36) questionnaire | 2 years
  SF-36 questionnaire in scores

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No